CLINICAL TRIAL: NCT04864925
Title: Measurement of Viral Load Reduction in the Oral Cavity After a Regimental Use of OC Toothpaste Products
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EXT-SARS2-COV2-OC-RUT-CD
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colgate Total Clean Mint (Experimental): Brush with toothpaste for a minimum of 2 minutes
  Interventions: Drug: Colgate Total Clean Mint
- Tom's Botanically Bright Peppermint (Active Comparator): Brush with toothpaste for a minimum of 2 minutes
  Interventions: Drug: Tom's Botanically Bright Peppermint

INTERVENTIONS:
Drug: Colgate Total Clean Mint — 2 minutes of whole mouth toothbrushing
  Other Names: Toothpaste
  Arms: Colgate Total Clean Mint
Drug: Tom's Botanically Bright Peppermint — 2 minutes of whole mouth toothbrushing
  Other Names: Toothpaste
  Arms: Tom's Botanically Bright Peppermint

SUMMARY:
SARS COVID 2 has caused a pandemic of proportions unparalleled in the past 100 years. The virus has an uncanny ability for transmission and as such has been difficult to control. The spread of the virus has affected everything from education, business, politics and survival. While the investigators have learned a great deal in the last 9 months they still face an uncertain day to day existence. Health care workers are particularly vulnerable to transmission of this virus because of their close contact with patients. Moreover, dentists are particularly vulnerable because the virus is spread via aerosols which are generated quite easily in the dental office putting dentists and their associates at risk. The oral cavity appears to be a likely domain for viral carriage particularly since both taste and smell are hallmark effects of the virus. With these issues at hand it will be of great advantage to have a simple routine oral hygiene method in the effort to reduce the oral viral load. There is some reason to expect that oral hygiene procedures with known anti-microbial effects could have some use in our efforts to reduce or control the oral viral load. With this issue in mind investigators feel that stannous fluoride could modify the virus in such a manner as to effectively reduce the oral viral load.

DETAILED DESCRIPTION:
Study will measure reduction of SARS-CoV-2 levels in the oral cavity after brushing for up to an hour. Subject sampling will occur at baseline, 15 min, 30 min, and 60 min

ELIGIBILITY:
Inclusion Criteria:

* Enrolled subjects between the ages of 18-64 and have tested positive for Covid19.

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR | Baseline
  Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR
Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR | 30 minutes after brushing
  Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR
Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR | 60 minutes after brushing
  Primary outcome based on reductions of viral titers in the oral cavity as determined by qRT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University Hospital, Newark, New Jersey, United States